CLINICAL TRIAL: NCT04623853
Title: Investigating Auto Adjusting Dynamic AFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joan Sanders, Professor: Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00009120
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lower Limb; Fusion, Congenital; Lower Limb Fracture; Ankle Foot Injury
Keywords: Ankle foot orthotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aim 2 (Experimental): Participants will carry out a protocol comprised of treadmill walking in a laboratory setting while wearing the Dynamic AFO device.
  Interventions: Device: Variable Stiffness AFO
- Aim 3 (Experimental): Participants will be asked to take the Dynamic AFO home and wear the device for up to 4 weeks. The device will be set in either an adjustment-capable mode, or a "locked" mode that functions similar to their own orthotic--the order in which they are tested will be randomized.
  Interventions: Device: Variable Stiffness AFO

INTERVENTIONS:
Device: Variable Stiffness AFO — The Dynamic AFO is able to adjust in stiffness depending on activity.

SUMMARY:
Offloading Ankle Foot Orthoses (AFOs) are devices designed for people following lower-limb reconstruction to restore mobility by reducing mechanical loading through the injury site and redistributing it proximally. While they perform well for some users, their current form limits full functional potential and may put joints proximal to the injury at risk of long-term damage. This study is directed toward designing and testing a lightweight, variable stiffness, dynamic brace that can adjust in response to user activity.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

-able to run continuously for 1 minute

Inclusion Criteria (All Other Volunteers)

* prescribed an offloading Ankle-Foot Orthosis (AFO) for walking/running
* Use prescribed offloading AFO at least 20 hours per week
* Prescribed AFO strut length of at least 200 mm
* Able to run continuously for 1 minute

Exclusion Criteria (Healthy Volunteers):

* limited sensation in the lower limbs
* use an assistive device

Exclusion Criteria (All Other Volunteers):

* Unable to ambulate (walk/run) continuously with AFO for at least 1 minute
* Unable to sit, stand, or negotiate a step onto lab treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time Running Per Day | Calculated across all days of data collection (up to 4 weeks).
  Collected while participant uses device in free-living environment.
Longest Running Bout Duration | Across all days of data collection (up to 4 weeks), the longest bout of continuous activity will be identified (minutes).
  Collected while participant uses device in free-living environment.
PROMIS-Fatigue | Following their time out in their free-living environment (up to 4 weeks at a time), participants will be asked to complete a questionnaire related to fatigue.
  Participants will be asked to fill out a questionnaire related to their experience using the variable stiffness AFO out of lab in various test configurations. Each PROMIS-Fatigue question asks participants to rank on a scale from 1 to 5 (categorical options), with higher scores indicating a greater level of fatigue.
Pain Score | Following their time out in their free-living environment (up to 4 weeks at a time), participants will be asked to complete a questionnaire related to pain.
  Participants will be asked to fill out a questionnaire related to their experience using the variable stiffness AFO out of lab in various test configurations. Each Pain-Score question asks participants to rank on a scale from 1 to 10 (categorical options), with higher scores indicating a greater level of pain.
Orthotic Evaluation Questionnaire (OEQ) | Following their time out in their free-living environment (up to 4 weeks at a time), participants will be asked to complete an OEQ.
  Similar to the Prosthesis Evaluation Questionnaire (PEQ), the OEQ will ask various questions concerning their experience wearing the variable stiffness AFO. Participants will rate their overall satisfaction, ability to ambulate, the health of their limb, the utility of the device, and their overall well-being after wearing the device.
Running Speed on Treadmill | In-lab testing will occur over the course of up to 2 hours at a time.
  Participants carrying out the in-lab protocol will be asked to run using the variable stiffness AFO and running speed will be documented at various time points.
Extended Figure-of-8 Test | In-lab testing wil occur over the course of up to 2 hours at a time.
  Participants carrying out the in-lab protocol will be asked to do a Figure-of-8 test.

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Sanders, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Dept. of Bioengineering, Seattle, Washington, United States